CLINICAL TRIAL: NCT05036005
Title: Neoadjuvant Treatment of Ontruzant (SB3) in Patients With HER2-positive Early Breast Cancer: An Open-Label, Multicenter, Phase IV Study
Brief Title: Neoadjuvant Ontruzant (SB3) in Patients With HER2-positive Early Breast Cancer: An Open-Label (NeoON)
Acronym: NeoON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut fuer Frauengesundheit (Other)
Collaborators: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFG-08-2019
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Female; HER2-positive Breast Cancer
Keywords: Ontruzant; Trastuzumab; Pertuzumab; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Ontruzant; Drug Therapy; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ontruzant + Pertuzumab (optional) + Chemotherapy (Experimental): All patients will receive 6 cycles of Ontruzant® i.v. q21d in combination with standard chemotherapy with or without pertuzumab, at the discretion of investigator's decision. Initial dose of Ontruzant® i.v. will be 8 mg/kg b.w. followed by 5 cycles of Ontruzant® i.v. 6 mg/kg b.w. q21d. Clinical and bioptic tumor assessment will be performed during baseline and during surgery.
  Study treatment will be applied until state of the art surgery, onset of unacceptable toxicities, progression or withdrawal of consent. A safety follow-up is planned for 30 days after the last administration of study medication.
  Interventions: Drug: Ontruzant; Drug: Chemotherapy; Drug: Pertuzumab

INTERVENTIONS:
Drug: Ontruzant — All patients will receive an initial dose of Ontruzant® i.v. 8 mg/kg b.w in combination with standard chemotherapy with or without pertuzumab i.v. 480 mg followed by 5 cycles of Ontruzant® i.v. 6 mg/kg b.w. q21d in combination with standard chemotherapy with or without pertuzumab i.v. 420 mg. Addition of pertuzumab is at the discretion of investigator's decision.
  Other Names: SB3
Drug: Chemotherapy — All patients will receive an initial dose of Ontruzant® i.v. 8 mg/kg b.w in combination with standard chemotherapy with or without pertuzumab i.v. 480 mg followed by 5 cycles of Ontruzant® i.v. 6 mg/kg b.w. q21d in combination with standard chemotherapy with or without pertuzumab i.v. 420 mg. Choice of chemotherapy is at the discretion of the investigator
Drug: Pertuzumab — All patients will receive an initial dose of Ontruzant® i.v. 8 mg/kg b.w in combination with standard chemotherapy with or without pertuzumab i.v. 480 mg followed by 5 cycles of Ontruzant® i.v. 6 mg/kg b.w. q21d in combination with standard chemotherapy with or without pertuzumab i.v. 420 mg. Addition of pertuzumab is at the discretion of investigator's decision.

SUMMARY:
The treatment of patients with HER2 positive early breast cancer has continuously improved over the last decades. Up to now both, trastuzumab and pertuzumab are approved in combination with chemotherapy (CTX) not only for the adjuvant but also for the neoadjuvant treatment of early breast cancer patients. A high pCR rate in the neoadjuvant setting was shown in several trials and observational studies with CTX+ trastuzumab and with CTX+ pertuzumab. The efficacy is dependent on a variety of mechanisms including the blocking of the important PI3K/Akt and MAPK pathways, and ADCC (antibody dependent cellular toxicity).

Recently the biosimilar Ontruzant® (SB3) has been introduced into the treatment of HER2 positive breast cancer as a biosimilar. Efficacy and toxicity have been shown to be equivalent to the first approved antibody, however, data from the real-world setting have not been published like it has for the originally approved antibody. Therefore, the aim of this study is to establish safety and efficacy for Ontruzant® in the real world setting. Patients can be included if they are treated with Ontruzant® in the neoadjuvant setting. Additionally, the study will be accompanied by a comprehensive immune monitoring program and biomarker program to explore immune oncology potential for the neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning of trial specific procedures.
2. Subject must be female and aged ≥ 18 years on day of signing informed consent.
3. ECOG 0-1.
4. Histologically confirmed, early HER2 positive breast cancer determined by core biopsy of breast tumor lesion.
5. Measurable tumor lesion with a size of ≥ 1 cm assessed by sonography or magnetic resonance imaging (MRI) within ≤ 28 days prior to entry. In case of inflammatory disease, the extent of inflammation will be measured.
6. Indication for chemotherapy.
7. Multicentric and/or multifocal disease as well as synchronous bilateral breast cancer is eligible as long as one measurable lesion meets all inclusion criteria. The investigator has to determine which lesion will be used for tumor evaluation before initiation of treatment.
8. Complete staging within 8 weeks prior to entry with no evidence of distant disease, including bilateral mammography, breast ultrasound, chest-X-ray (or chest CT-scan), liver ultrasound (or liver CT-scan or liver MRI) and bone scan.
9. Subjects must provide a core biopsy from tumor lesion before first chemotherapy, after 3 cycles of chemotherapy and after last neoadjuvant study treatment for biomarker analyses.
10. Adequate organ function defined as: Absolute neutrophile count ≥1500/µL, Platelets ≥100 000/µL, Hemoglobin ≥10.0 g/dL or ≥6.2 mmol/L, Creatinine ≤1.5 × ULN OR measured or calculated creatinine clearance ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN (GFR can also be used in place of creatinine or CrCl), Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN, AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases), International normalized ratio (INR) OR prothrombin time (PT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants, LVEF > 50 %
11. Female subjects of childbearing potential must have a negative urine pregnancy test within 72 h prior to study entry and be willing to use an adequate method of contraception for course of the study through 7 months after the last dose of trial treatment.

Exclusion Criteria:

1. Concurrent participation in a study with an investigational agent/device or within 14 days of study entry.
2. Prior chemotherapy, radiation therapy or small molecule therapy for any reason.
3. Previous malignant disease being disease-free for less than 3 years (except in situ carcinoma of the cervix and basal cell carcinoma of the skin).
4. Pregnancy or lactation.
5. Prior neoadjuvant therapy.
6. Active infection requiring systemic therapy.
7. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
8. Active autoimmune disease or other diseases that requires systemic treatment with corticosteroids or immunosuppressive drugs (physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is allowed).
9. History of primary or acquired immunodeficiency (including allogenic organ transplant).
10. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
11. Known history of following infections: Human immunodeficiency virus (HIV), History of acute or chronic Hepatitis B or Hepatitis C, has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
12. Known congestive heart failure > NYHA I and/or coronary heart disease, angina pectoris, previous history of myocardial infarction, uncontrolled or poorly controlled arterial hypertension (e.g. blood pressure >160/90 mmHg under treatment with two or more antihypertensive drugs), rhythm disorders with clinically significant valvular heart disease.
13. Pre-existing motor or sensory neuropathy of a severity grade ≥2 by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
14. Any other condition in opinion of the investigator that would interfere with applied systemic treatment or other trial procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-07-11 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Pathological complete response will be assessed at final surgery.
  Pathological complete response (pCR) rate, defined as the complete absence of tumor cells (ypT0; ypN0) after neoadjuvant study treatment of HER2-positive early breast cancer patients treated with Ontruzant® (SB3) in combination with pertuzumab (optional) and a standard chemotherapy.

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate in patients without pertuzumab | Pathological complete response will be assessed at final surgery.
  Pathological complete response (pCR) rate, defined as the complete absence of tumor cells (ypT0; ypN0) after neoadjuvant study treatment of HER2-positive early breast cancer patients treated with Ontruzant® (SB3) and a standard chemotherapy who were not treated with pertuzumab.
Number of participants wuth treatment-related adverse events as assessed by CTCAE v5.0 | Adverse ebents will be assessed from first administration of trial treatment until 30 days after last administration of trial treatment.
  The safety endpoints for the study will include rate of AE/SAEs and fatal SAEs, causality and outcome of AE/SAEs, rate of treatment discontinuations and reasons, Changes in vital signs, laboratory values etc. Grading of AE/SAEs will be based on NCI CTCAE v5.0.
EORTC-QLQ-C30 | Every nine weeks from first administration of trial medication through study completion, up to 30 days after administration of last medication.
  To evaluate changes in health related quality of life (QoL) assessments from baseline in all subjects using Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
EORTC-QLQ-BR23 | Every nine weeks from first administration of trial medication through study completion, up to 30 days after administration of last medication.
  To evaluate changes in health related quality of life (QoL) assessments from baseline in all subjects using Quality of Life Questionnaire Breast Cancer-Specific Quality of Life (EORTC QLQ-BR23).

OTHER OUTCOMES:
To assess the antibody-dependent cell mediated cytotoxicity (ADCC) | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery
  ADCC will be quantified and immune phenotyping will be performed from peripheral blood mononuclear cells (PBMCs).
FcγR genotypes | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery
  Germline DNA will be genotyped in order to specify FcγR polymorphisms and impact of FcγR genotypes on ADCC and pCR will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Lüftner, MD, Prof., Study Chair — Department for Hematology, Oncology and Tumor Immunology Charité Campus Benjamin Franklin, Berlin; Andreas Schneeweiss, MD, Prof., Study Chair — National Center for Tumor Diseases (NCT), Head of Division Head of Division Gynecologic Oncology, Heidelberg University Hospital (UKHD)
Locations (11):
- Germany (11):
  - Division Gynecologic Oncology, Heidelberg University Hospital (UKHD), Heidelberg, Baden-Wurttemberg
  - Department of Gynecology, Tübingen University Hospital, Tübingen, Baden-Wurttemberg
  - Hämato-Onkologische Schwerpunktpraxis am Klinikum Aschaffenburg, Aschaffenburg, Bavaria
  - Department of Gynecology and Obstetrics, Erlangen University Hospital, Erlangen, Bavaria
  - Department of Gynecology, University Hospital Hamburg-Eppendorf, Hamburg, Haburg
  - Center for Hematology and Oncology Bethanien, Frankfurt am Main, Hesse
  - Department of Gynecology and Obstetrics, University Medicine Mainz, Mainz, Hesse
  - Department for Gynecology and Obstetrics, Marienhospital Bottrop gGmbH, Bottrop, North Rhine-Westphalia
  - Department of Gynecology and Obstetrics, Dresden University Hospital Carl-Gustav Carus, Dresden, Saxony
  - Department for Hematology, Oncology and Tumor Immunology Charité Campus Benjamin Franklin, Berlin
  - Department of Gynecology and Obstetrics, HELIOS Hospital Berlin Buch GmbH, Berlin

IPD SHARING:
Plan to Share IPD: No